CLINICAL TRIAL: NCT01519336
Title: A Study to Evaluate the Potential Drug-Drug Interaction Between Darunavir and Danoprevir When Administered Together With Low-Dose Ritonavir in Healthy Volunteers
Brief Title: A Study of Drug-Drug Interaction Between Darunavir and Danoprevir Administered Together With Low-Dose Ritonavir in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: NP28089
Record Dates: First submitted 2012-01-24; First posted 2012-01-26 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — danoprevir; Darunavir; Ritonavir

ARMS (3):
- A danoprevir (Active Comparator)
  Interventions: Drug: danoprevir; Drug: ritonavir
- B darunavir (Placebo Comparator)
  Interventions: Drug: darunavir; Drug: ritonavir
- C danoprevir/darunavir (Experimental)
  Interventions: Drug: danoprevir; Drug: darunavir; Drug: ritonavir

INTERVENTIONS:
Drug: danoprevir — 100 mg q12h
  Arms: A danoprevir; C danoprevir/darunavir
Drug: darunavir — 600 mg q12h
  Arms: B darunavir; C danoprevir/darunavir
Drug: ritonavir — 100 mg q12h

SUMMARY:
This randomized, open-label, multiple-dose, 2-period crossover study will evaluate potential drug-drug interactions between darunavir and danoprevir when administered together with low-dose ritonavir in healthy volunteers. In Period 1, subjects will be randomized to receive either darunavir or danoprevir together with low-dose ritonavir for 10 days. In Period 2, all subjects will receive darunavir plus danoprevir together with ritonavir for 10 days. Anticipated time on study treatment is 20 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking male and female adults, 18 - 55 years of age, inclusive
* Healthy status defined by absence of evidence of any active or chronic disease
* Medical history without major, recent, or ongoing pathology
* Weight >/= 55 kg
* Body mass index (BMI) 18.0 - 32.0 kg/m2
* Ability and willingness to abstain from alcohol, xanthine-containing beverages or food (coffee, tea, cola, chocolate, "energy drinks") from 72 hours prior to entry in the clinical site center until discharge
* Females of child-bearing potential and males and their female partners of child-bearing potential must agree to use 2 forms of contraception, one of which must be a barrier method, during the study and for 90 days after the last drug administration. Acceptable barrier forms of contraception are condom and diaphragm; acceptable non-barrier forms of contraception for this study are non-hormonal intrauterine device (IUD) and/or spermicide

Exclusion Criteria:

* Pregnant or lactating females or males with female partners who are pregnant or lactating
* Any history of clinically significant cardiovascular or cerebrovascular disease, hypertension, and/or infections
* Positive test for drugs of abuse at screening or prior to admission to the clinical site during any study period
* Positive for hepatitis B, hepatitis C or HIV infection
* Current smokers or subjects who have discontinued smoking less than 6 months prior to first dose of study medication
* Use of hormonal contraceptives within 30 days before the first dose of study medication
* History of clinically significant drug-related allergy (such as anaphylaxis) or hepatotoxicity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Effect of coadministration of darunavir (DRV), danoprevir (DNV) and ritonavir (RTV) on DRV/DNV/RTV pharmacokinetics: Area under the concentration-time curve (AUC) | approximately 2 months

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Lenexa, Kansas, United States